CLINICAL TRIAL: NCT03606525
Title: Correlation Between Vertebral Column Length (VCL), Abdominal Circumference (AC) and Spread of Intrathecal Hyperbaric Bupivacaine in the Term Parturient
Brief Title: Correlation Between VCL, AC and Spread of Intrathecal Hyperbaric Bupivacaine in the Term Parturient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Soo Suet Ker, Medical officer, Department of Anaesthesiology, Principal investigator, University of Malaya
Other Study IDs: 201843-6195
Record Dates: First submitted 2018-07-02; First posted 2018-07-31 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Effects of; Anesthesia, Spinal and Epidural, in Pregnancy
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: subarachnoid block — Vertebral column length and abdominal girth will be measured before routine subarachnoid block is given to recruited patients

SUMMARY:
Currently there is no guideline to decide on the most appropriate dose of spinal anaesthesia. This study is planned to find out factors that influence the effect of spinal anaesthesia in pregnant mother going for Caesarean section and both the mother and baby's outcomes. Investigators will recruit pregnant mothers who are planned for elective Caesarean section under spinal anaesthesia at University Malaya Medical Centre before operation and obtained their consent to participate in this study. Routine standard care will be provided for all the participants. Perioperative data including vertebral column length and abdominal girth measured by measuring tape will be collected and analysed. There is no new intervention performed on participants.

DETAILED DESCRIPTION:
The rising rate of caesarean section is a global phenomenon. Rate of caesarean section in Malaysia were 23.41% in 2011 and 25.08% in 2012. Subarachnoid block is the preferred anaesthetic technique for most lower segment caesarean section as compared to general anaesthesia. This is because general anaesthesia is associated with higher risk of failed endotracheal intubation and aspiration of gastric contents in parturients. Moreover, usage of pencil-point spinal needle had reduced the risk of postdural puncture headache frequency and severity.

Effective surgical anaesthesia is the main objective of subarachnoid block. Therefore, adequate sensory blockade with minimal maternal and neonate side effects are warranted. The suitable level of sensory blockade post subarachnoid block for lower segment caesarean section is bilateral block up to T6 dermatome level to pinprick. This will block the somatic sensation and eliminate the visceral pain from peritoneal manipulation during caesarean section.

However, the spread of subarachnoid block may be variable. Various patient variables such as age, height, weight, body mass index, vertebral column length and abdominal girth influence the spread of subarachnoid block. Inadequate sensory blockade will cause parturient suffer from pain while excessive blockade will lead to unwanted sympathetic inhibition causing hypotension and bradycardia. Ability of an anaesthetist to determine optimal dose to achieve adequate level of sensory blockade yet with minimal unwanted side effects is crucial.

Incidence of maternal hypotension is related to the level of sensory blockade after subarachnoid block.And maternal hypotension is associated with maternal discomfort during caesarean section and poorer fetal outcomes. Therefore, this study is carried out to investigate whether vertebral column length and abdominal circumference affecting the spread of intrathecal hyperbaric bupivacaine in term parturient.

Previous studies showed conflicting results on the factors that influence the effect of spinal anaesthesia. One of the studies was carried out in China which might not reflect the investigator's local multiracial population characteristics. Previous studies also did not investigate the outcome of baby related to maternal hypotension which is known complication.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 18 years old
* American Society of Anesthesiologists (ASA) physical status I-II
* singleton pregnancy
* gestational age 37 weeks or more
* height 150-175cm and weight 50-100kg

Exclusion Criteria:

* patients with contraindication to subarachnoid block
* history of allergy to local anaesthetics
* contraindication to NSAIDS use
* failure of subarachnoid block
* any abnormality of spine
* history of spinal surgery
* refusal to participate in this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all term parturients going for elective Caesarean section
Study Population: term parturients who are scheduled for elective Caesarean section under spinal anaesthesia in University Malaya Medical Centre
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
sensory block level | 15 minutes after subarachnoid injection
  Pin-prick test will be performed in both midclavicular lines to determine to level of sensory blockade every 3 minutes. Highest level of sensory blockade will record at 15 minutes after intrathecal injection.

SECONDARY OUTCOMES:
blood pressure post subarachnoid block | 2 hours
  Both systolic and diastolic blood pressure will be taken every 5 minutes until Caesarean section is completed
regression of subarachnoid block | 1day
  Motor block will be assessed every hour until complete motor recovery or 6 hours after subarachnoid block, according to modified Bromage scale (Breen et al) as follows: 1= complete block (unable to move feet or knees); 2= almost complete block (able to move feet only); 3= partial block (just able to move knees); 4= detectable weakness of hip flexion while supine (full flexion of knees); 5= no detectable weakness of hip flexion while supine; 6= able to perform partial knee bend while assume standing position.

CONTACTS AND LOCATIONS:
Overall Officials: Suet Ker Soo, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou QH, Xiao WP, Shen YY. Abdominal girth, vertebral column length, and spread of spinal anesthesia in 30 minutes after plain bupivacaine 5 mg/mL. Anesth Analg. 2014 Jul;119(1):203-206. doi: 10.1213/ANE.0000000000000199. PMID 24806139
- [Background] Zhou QH, Zhu B, Wei CN, Yan M. Abdominal girth and vertebral column length can adjust spinal anesthesia for lower limb surgery, a prospective, observational study. BMC Anesthesiol. 2016 Mar 24;16:22. doi: 10.1186/s12871-016-0184-3. PMID 27009023